CLINICAL TRIAL: NCT06364969
Title: Investigation of the Pruritogens of Liver-related Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-06-02
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Cholestasis; Intrahepatic Cholestasis of Pregnancy
Keywords: cholestasis; pruritus
MeSH Terms: conditions — Cholestasis; Intrahepatic Cholestasis of Pregnancy; Pruritus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy subjects: Healthy adult volunteers (aged 18-35 years)

SUMMARY:
This study hopes investigate the itch-inducing ability of different potential pruritogen candidates of cholestasis pruritus, especially the intrahepatic cholestasis of pregnancy (ICP). In this study, a combination of skin application and needle-free subcutaneous injection was used to investigate whether human endogenous molecules can cause itching. And a questionnaire is used to quantify the intensity of different candidates-induced itch.

DETAILED DESCRIPTION:
Liver-related diseases are a large group of diseases that seriously affect people's healthy life. For example, ICP, the most common liver-related disease in pregnancy, affects on average about 4% of pregnant women worldwide. In a cohort study of 12200 eligible Chinese pregnant women, the reported incidence of ICP was 6.06%. ICP is harmful to the health of both pregnant women and fetuses. For the fetus, ICP directly affects the healthy growth and smooth delivery of the fetus. Disease-related adverse events have been reported, including preterm birth, meconium contamination of amniotic fluid, fetal hypoxia, prolonged length of stay in neonatal unit, and even stillbirth. ICP has a serious impact on the physical and mental health of pregnant women, typically severe pruritus. This itching occurs mainly in the second and third trimesters of pregnancy (usually the third trimester) and tends to become progressively worse as the pregnancy progresses. It is most commonly present on the palms and soles of the feet, and some patients have generalized itching. Moreover, the itching was aggravated at night, leading to severe insomnia. Under the background of advocating multiple births in our country, the effective prevention and treatment of such diseases is particularly important.

At present, there are no effective drugs for the treatment of ICP, especially pruritus symptoms, because the molecular mechanism of ICP and its pruritus is still unclear. In this study, we have identified several endogenous potential pruritogens that can activate human MRGPRX4 (hX4), the potential itch receptor of ICP pruritus, to mediate ICP pruritus based on a large number of previous cell and animal experiments. On this basis, the present study aims to evaluate the direct pruritic ability of different endogenous metabolites through human psychophysical experiments and subcutaneous administration of drugs to human subjects through a needle-free injection system.

In detail, this study includes two parts.

1. Test whether the molecule causes itching i) Skin application: a certain amount of human endogenous metabolites (progesterone sulfates) are dissolved in Cold cream (Avene, France). Firstly, disposable medical disinfection cotton (Lu Qing Food and Drug Supervision and Equipment (Zhun) word 2013 No. 1640069) is used to disinfect the forearm flexor skin of healthy adult subjects. The cream is then applied to the surface of the forearm (double-blind requirements were followed). During the experiment, the subjects complete the itch and pain perception questionnaire. At the end of the experiment, the changes in the administration area are observed and recorded by the chief test, including whether erythema and wheals occur.

   ii) Needle-free subcutaneous injection: a certain amount of human endogenous metabolites or FDA-approved drugs is dissolved in normal saline. Firstly, disposable medical disinfection cotton (Lu Qing Food and Drug Supervision and Equipment (Zhun) word 2013 No. 1640069) is used to disinfect the forearm skin of healthy adult subjects. Then, the drug solution is injected into the forearm surface of healthy adults using the clinical insulin injection needle-free injection system (INJEX30 needle-free injection system) (China Food and Drug Supervision Instrument (Jin) Word 2013 No. 3151260). The system mainly includes a disposable syringe, a pressurizer, a disposable ampoule and a disposable shock cushion. During the experiment, the subjects complete the itch and pain perception questionnaire. At the end of the experiment, the changes in the administration area are observed and recorded by the chief test, including whether erythema and wheals occur.
2. Molecular mechanisms of pruritus About 2g antihistamine cream (doxepin hydrochloride cream, H20041591) and placebo (Cold cream, Avene, France) are applied to the flexor muscles of the forearm (about 4cm2). After 2 hours, the drug is administered as a skin application or needle-free subcutaneous injection as described above: 2.5ug of histamine (positive control) and the indicated doses of the aforementioned potentially itch-causing molecule (double-blind requirements were followed). The changes of the skin administration area (whether there is erythema and wheals) are observed during the experiment, and the subjects complete the itch and pain perception questionnaires.
3. Psychophysical experiments The general Labeled Magnitude Scale (gLMS) is used to estimate the level of itch (or pain) at the current moment, relative to the level of itch (or pain) experienced by the subjects in previous situations. Subjects chose from the following adjectives to describe the degree of itching (or pain) : ① barely felt, ② faint, ③ mild, ④ intense, ⑤ very intense, or ⑥ most intense.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers

Exclusion Criteria:

* People with mental disorders, bone or skeletal muscle disorders, psychological disorders, various skin diseases, allergic symptoms, and similar medical histories
* People with itching or pain symptoms
* People who were on medication

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Both male and female Healthy adult volunteers (aged 18-35 years)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Itch intensity | Half an hour after receiving the injection
  by questionnaire

SECONDARY OUTCOMES:
Flare areas | Half an hour after receiving the injection
  Measuring by the ruler

CONTACTS AND LOCATIONS:
Overall Officials: Yulong Li, Principal Investigator — Peking University
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Privacy and competition

REFERENCES:
- [Background] Yu H, Zhao T, Liu S, Wu Q, Johnson O, Wu Z, Zhuang Z, Shi Y, Peng L, He R, Yang Y, Sun J, Wang X, Xu H, Zeng Z, Zou P, Lei X, Luo W, Li Y. MRGPRX4 is a bile acid receptor for human cholestatic itch. Elife. 2019 Sep 10;8:e48431. doi: 10.7554/eLife.48431. PMID 31500698